CLINICAL TRIAL: NCT04638842
Title: Effectiveness of a Self-applied Multi-component Psychological Online Intervention Based on UX, for the Prevention of Complicated Grief Disorder in the Mexican Population During the COVID-19 Outbreak: A Randomized Clinical Trial
Brief Title: Online Multi-component Psychological Intervention for Prevention of Grief Disorder Due to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Internacional de Valencia (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); Universidad Autonoma de Ciudad Juarez (Other); University of Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIU-Grief-COVID
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Grief; Anxiety; Depression; Sleep Disturbance; Quality of Life
MeSH Terms: conditions — Anxiety Disorders; Depression; Parasomnias

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the experimental group that receives the treatment and the other is the comparison group that will receive treatment after the 12 sessions of the experimental group finished. The patients in both groups will be evaluated pre and post/treatment. The participants are assigned randomly to the intervention or comparison group.
Who Masked: Participant
Masking Description: The patients are not aware that there is an experimental group and a control group, the participants are not related and do not know each other. The conditions of the study are only known by the researcher, the therapists, and the Research Ethics Committee of the Universidad Autónoma de Ciudad Juárez.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grief COVID intervention (Experimental): Participants in this group will receive 12 sessions of a multi-component psychological intervention focused on the reduction of symptoms of anxiety, depression, hopelessness, and post-traumatic stress, and the increase of the quality of sleep and perception of the quality of life.
  Interventions: Behavioral: Online Intervention Grief COVID-19
- Waiting List group (No Intervention): The participants in this group will not receive the treatment, just waiting list. They will be measured one time and then a second time 3 months after. Calculating when 3 months corresponding to 12 sessions will receive the intervention.

INTERVENTIONS:
Behavioral: Online Intervention Grief COVID-19 — The online Intervention Grief COVID-19 aims to provide to the target population a self-applied intervention based on Cognitive Behavioral Therapy, Mindfulness, Behavioral Activation Therapy, and Positive Psychology, aimed at the Psychoeducation regarding the manifestations of normal grief, advice and guidance on how to find emotional relief, with the aim that survivors allow themselves to validate their experience of emotional pain and recognize it as a normal part of their process of adaptation to loss, what does grief deprived of rights consist of, specifically from the contingency of COVID-19, establish self-care measures for people in different areas of their life (physical, emotional, cognitive and spiritual), direct the survivor to relocate the died in his life without his memory causing suffering, in addition to beginning to resume his life project, adjusting according to his needs and goals. The sessions will be delivered in a frequency of one session every three days.
  Arms: Grief COVID intervention

SUMMARY:
This study evaluates the effectiveness of an online Multi-component psychological intervention, that is focused on providing self-support to the Mexican population for the prevention of complicated grief disorder, by reducing grief and strengthening the capacities of the person to handle losses derived from COVID-19 as well as reducing the symptoms of anxiety, depression, hopelessness, and post-traumatic stress, and increasing the quality of sleep and perception of the quality of life.

DETAILED DESCRIPTION:
The loss of a loved one is perhaps one of the most shocking events in the life of a person. Grief is an emotional experience universal human, unique and painful, that can be delimited in time, which allows the person to adapt to loss and the new reality. In situations, prior to COVID-19, there was a risk of suffering prolonged grief when going through the death of a family member hospitalized and unable to say goodbye. The global COVID-19 pandemic is expected to have a major impact related to the experience of death, dying, and grief, which will make the grieving process difficult. The confusion, anger, and post-traumatic stress are some of the negative effects related to quarantine. It is not only difficult to deal with the loss of the person but at the same time with the interruption of rituals and practices associated with a death such as funerals and burials, which are postponed and performed without the presence of family. Given such data, it is necessary to intervene with proposals that help improve mental health and the management of grief.

To provide treatment in such conditions where face-to-face sessions are not possible, and the number of patients surpasses the number of available therapists it will be implemented an online intervention based on Cognitive Behavioral Therapy, Mindfulness, Behavioral Activation Therapy, and Positive Psychology. The Online Intervention system "Grief COVID" will be delivered in 12 modules interconnected. The objective of this study is to assess the efficacy and moderators of change of this intervention for the reduction of symptoms of anxiety, depression, hopelessness, and post-traumatic stress, and the increase of the quality of sleep and perception of the quality of life.

The contents of this intervention will be implemented through a responsive web application. In order to create the most fitted intervention for the real needs of the participants will be created following the principles of User Experience (UX), with this ensuring that the design characteristics of the tool will meet the desired requirements to be perceived as easy to use, attractive and useful. The UX approach refers to the experience that a user has with a product, with special emphasis on human-product interaction.

This study will have an experimental and control group. The experimental group will receive the intervention to prevent complicated grief, and the control group will be on the waiting list. Participants will be randomly assigned to one of the two groups. Participants in the control group once their data have been collected and the time elapsed after receiving the intervention in the participants in the experimental group will receive access to the intervention and will also be evaluated in order to increase the sample level and to be able to have more results about the effectiveness of the intervention. In both conditions, the participants will be measured at pre and post moments. The subjective measures will include the following Psychometrics:

1. Depression scale of the Center for Epidemiological Studies.
2. The abbreviated depression, anxiety, and stress scale (DASS-21).
3. Plutchik Suicide Risk Scale.
4. Pittsburgh Sleep Quality Index.
5. Post-traumatic diagnostic scale.
6. Satisfaction with Life Scale.
7. Beck's Hopelessness Scale.
8. Generalized Anxiety Scale (GAD-7).
9. Opinion on the treatment.
10. System usability scale.

ELIGIBILITY:
Inclusion Criteria:

* To have access to a communication device with access to the internet (computer, tablet, and mobile).
* To have a valid email address.
* To have basic digital skills in the use of an operational system and internet browsing.
* To understand Spanish since all the contents are in this language.
* Having suffered the loss of a loved one in a period of no less than 3 months and no longer than 6 months.
* Symptoms of General Anxiety Disorder and/or Depression and/or, grief symptoms.

Exclusion Criteria:

* To have a diagnosis of psychotic disorder
* To be receiving psychological and/or pharmacological treatment during the study
* Moderate to high score on the suicide scale
* Recent attempt of suicide (3 months)
* Symptoms of posttraumatic Stress Disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Decrease in the scores of the Center for Epidemiologic Studies Depression (CES-D) scale | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  Center for Epidemiologic Studies Depression (CES-D) is a structured self-report scale for evaluation depression symptoms. This scale assesses the number of depression symptoms within 2 weeks. The scale consists 20 items and contains 4-point score responses (0 to 3) as the following; rarely or none of the time (less than 1 day); some of a little of the time (1-2 days); occasionally or moderate amount of time (3-4 days) and most or all of the time (5-7 days). The total possible range of scores is from 0 to 60 where ^16 is the cut-off point for this scale, and higher scores indicate more symptoms of depression. It is expected a statistically significant decrease (P < 0.05) in depression symptoms.
Change in the score of Anxiety Symptoms in the Depression Anxiety Stress Scale (DASS-21) | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  The Depression Anxiety Stress Scale-21 is a structured self-report scale that assesses the subscales of anxiety, depression, and stress symptoms over the past last week. Each subscale contains seven items with responses rated on a 4-point scale (0-3) as follows; 0 Did not apply at me at all; 1 Applied to me to a considerable degree or some of the time; 2 Applied to me to a considerable degree or a good part of the time; 3 Applied to me very much or most of the time. Each subscale has a cut-off point for depression (6), anxiety (5), and stress (6). It is expected a statistically significant decrease (P < 0.05) in depression and anxiety symptoms.
Decrease in the score of The Pittsburgh Sleep Quality Index. | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  This instrument assesses the quality patterns of sleep. It differentiates the "poor" and "good" sleep by measuring seven areas, where the range score of answers are from 0 to 3, the global sum of this scale can be a value between 0 to 60, and the cutoff point is "5" that indicates a "poor" sleep quality. It is expected a statistically significant increase (P < 0.05) in the Sleep Quality measure.
Decrease in the scores of the Post-Traumatic Stress Disorder Symptom Scale | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  The Post-Traumatic Stress Disorder Symptom Scale is a 17-item structured interview. The severity over the last 2 weeks of each item on the PSS is rated by the interviewer using a 4-point scale: 0 = not at all, 1 = a little bit, 2 = somewhat, and 3 = very much. The maximum possible score is 51 (severely affected) and the minimum possible score is 0 (total absence of the symptoms). The total severity score is calculated as the sum of the severity ratings for the 17 items. The diagnosis of the Post-Traumatic Stress Disorder Symptom Scale is made when at least 1 re-experiencing, 3 avoidance, and 2 arousal symptoms are endorsed on the scale by individuals who were traumatized at least one month prior to the assessment. It is expected a statistically significant decrease (P < 0.05) in the symptoms of Post-Traumatic Stress Disorder in the patients suffering from this disorder.
Increase in Satisfaction with Life Scale | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  This instrument is composed of 5 items in which the participants must indicate how much they agree with each question, with an answer option in Likert format from 1 (totally disagree) to 7 (totally agree), the scores range from a minimum from 5 to a maximum of 35, where the highest scores indicate greater satisfaction with life. This scale has been validated in the Mexican population, obtaining good results of internal consistency (α = 0.74).
Decrease in the symptoms of General Anxiety Disorder | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  On the Generalized Anxiety Disorder 7-item (GAD-7) scale subjects are asked how often, during the last 2 weeks, they have been bothered by each of the 7 core symptoms of generalized anxiety disorder. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of ≥5, ≥10, and ≥15 represent mild, moderate, and severe anxiety symptom levels, respectively. Is expected a statistically significant decrease (P < 0.05) in the General Anxiety symptoms.

SECONDARY OUTCOMES:
Decrease in the Plutchik Suicide Risk Scale | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  The Plutchik Suicide Risk Scale is a structured self-report questionnaire for evaluating Suicide Risk. It consists of 15 items that assess the history of suicide attempts, ideation, and suicide plans. It differentiates patients with a suicide risk from the non-suicide risk. This scale has dichotomous responses of Yes/No, and has a cut-off point of 6, where a point above the cut-off means a higher suicide risk. In this study, the suicidal patients are not considering the depression treatment although is necessary to assess depressive patients to refer to specialized treatment.
Decrease in Grief symptoms | 1.5 to 2 months, depending on the development of the patient and the completion of the 12 modules
  The inventory of Complicated Grief is composed of 19 items, with a five Likert-type scale ranging from 0 to 4, where: 0 "never", 1 "rarely, 2" sometimes ", 3" often "and 4" always ". The items assess the frequency of the explored symptoms type (emotional, cognitive or behavioral). For its evaluation, the points of each item are added and the scores fluctuate between 0 and 76 points, scores above 25 are an indicator of complicated grief.

CONTACTS AND LOCATIONS:
Overall Officials: Sofía Cristina Martínez Luna, MD, Study Chair — Universidad Nacional Autonoma de Mexico; Paulina Arenas Landgrave, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Anabel de la Rosa, Gómez, Study Chair — Universidad Nacional Autonoma de Mexico; Esteban Eugenio Esquivel Santoveña, PhD, Study Chair — Universidad Autónoma de Ciudad Juárez; Rosa Olimpia Castellanos Vargas, MD, Study Chair — Universidad Autónoma de Ciudad Juárez; Luis Farfallini, PhD, Study Chair — University of Buenos Aires
Locations (1):
- Universidad Autónoma de Ciudad Juárez, Juárez, Chihuahua, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, ICF
Time Frame: This data will be available approximately in April 2021 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Wallace CL, Wladkowski SP, Gibson A, White P. Grief During the COVID-19 Pandemic: Considerations for Palliative Care Providers. J Pain Symptom Manage. 2020 Jul;60(1):e70-e76. doi: 10.1016/j.jpainsymman.2020.04.012. Epub 2020 Apr 13. PMID 32298748
- [Background] Holland DE, Vanderboom CE, Dose AM, Moore D, Robinson KV, Wild E, Stiles C, Ingram C, Mandrekar J, Borah B, Taylor E, Griffin JM. Death and Grieving for Family Caregivers of Loved Ones With Life-Limiting Illnesses in the Era of COVID-19: Considerations for Case Managers. Prof Case Manag. 2021 Mar-Apr 01;26(2):53-61. doi: 10.1097/NCM.0000000000000485. PMID 33181608
- [Background] Mayland CR, Harding AJE, Preston N, Payne S. Supporting Adults Bereaved Through COVID-19: A Rapid Review of the Impact of Previous Pandemics on Grief and Bereavement. J Pain Symptom Manage. 2020 Aug;60(2):e33-e39. doi: 10.1016/j.jpainsymman.2020.05.012. Epub 2020 May 15. PMID 32416233
- [Background] Boelen PA, Prigerson HG. The influence of symptoms of prolonged grief disorder, depression, and anxiety on quality of life among bereaved adults: a prospective study. Eur Arch Psychiatry Clin Neurosci. 2007 Dec;257(8):444-52. doi: 10.1007/s00406-007-0744-0. PMID 17629728
- [Background] Boelen PA, Smid GE. Disturbed grief: prolonged grief disorder and persistent complex bereavement disorder. BMJ. 2017 May 18;357:j2016. doi: 10.1136/bmj.j2016. No abstract available. PMID 28522468
- [Background] Sauer J, Sonderegger A, Schmutz S. Usability, user experience and accessibility: towards an integrative model. Ergonomics. 2020 Oct;63(10):1207-1220. doi: 10.1080/00140139.2020.1774080. Epub 2020 Jun 12. PMID 32450782
- [Background] Merino MD, Privado J. Positive Psychological Functioning. Evidence for a new construct and its measurement.[Funcionamiento psicológico positivo. Evidencia para un nuevo constructo y su medición]. Anales de Psicología/Annals of Psychology. 2015;31(1):45-54.
- [Background] Foa EB, Cashman L, Jaycox L, Perry K. The validation of a self-report measure of posttraumatic stress disorder: the Posttraumatic Diagnostic Scale. Psychological assessment. 1997 Dec;9(4):445.
- [Background] Kersting A, Dolemeyer R, Steinig J, Walter F, Kroker K, Baust K, Wagner B. Brief Internet-based intervention reduces posttraumatic stress and prolonged grief in parents after the loss of a child during pregnancy: a randomized controlled trial. Psychother Psychosom. 2013;82(6):372-81. doi: 10.1159/000348713. Epub 2013 Sep 20. PMID 24061387
- [Background] Hoffmann R, Grosse J, Nagl M, Niederwieser D, Mehnert A, Kersting A. Internet-based grief therapy for bereaved individuals after loss due to Haematological cancer: study protocol of a randomized controlled trial. BMC Psychiatry. 2018 Feb 27;18(1):52. doi: 10.1186/s12888-018-1633-y. PMID 29482525
- [Background] Sogaard Neilsen A, Wilson RL. Combining e-mental health intervention development with human computer interaction (HCI) design to enhance technology-facilitated recovery for people with depression and/or anxiety conditions: An integrative literature review. Int J Ment Health Nurs. 2019 Feb;28(1):22-39. doi: 10.1111/inm.12527. Epub 2018 Aug 22. PMID 30133096
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Carleton RN, Thibodeau MA, Teale MJ, Welch PG, Abrams MP, Robinson T, Asmundson GJ. The center for epidemiologic studies depression scale: a review with a theoretical and empirical examination of item content and factor structure. PLoS One. 2013;8(3):e58067. doi: 10.1371/journal.pone.0058067. Epub 2013 Mar 1. PMID 23469262
- [Result] Norton PJ. Depression Anxiety and Stress Scales (DASS-21): psychometric analysis across four racial groups. Anxiety Stress Coping. 2007 Sep;20(3):253-65. doi: 10.1080/10615800701309279. PMID 17999228
- [Result] Koslowsky M, Bleich A, Greenspoon A, Wagner B, Apter A, Solomon Z. Assessing the validity of the Plutchik Suicide Risk Scale. J Psychiatr Res. 1991;25(4):155-8. doi: 10.1016/0022-3956(91)90019-7. PMID 1779413
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Result] Novy DM, Stanley MA, Averill P, Daza P. Psychometric comparability of English- and Spanish-language measures of anxiety and related affective symptoms. Psychol Assess. 2001 Sep;13(3):347-55. doi: 10.1037//1040-3590.13.3.347. PMID 11556271
- [Derived] Dominguez-Rodriguez A, Sanz-Gomez S, Gonzalez Ramirez LP, Herdoiza-Arroyo PE, Trevino Garcia LE, de la Rosa-Gomez A, Gonzalez-Cantero JO, Macias-Aguinaga V, Miaja M. The Efficacy and Usability of an Unguided Web-Based Grief Intervention for Adults Who Lost a Loved One During the COVID-19 Pandemic: Randomized Controlled Trial. J Med Internet Res. 2023 Apr 6;25:e43839. doi: 10.2196/43839. PMID 36877800

DOCUMENTS (1):
  • Informed Consent Form (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04638842/ICF_000.pdf